CLINICAL TRIAL: NCT03706417
Title: Leveraging Telemedicine to Reduce Disparities in Time to Initiation of Therapeutic Hypothermia in Rural Settings; a Pilot Feasibility Study
Brief Title: Telemedicine to Improve Use of Therapeutic Hypothermia in Rural Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MaineHealth (Other)
Responsible Party: Principal Investigator, Alexa Craig, Associate Professor of Pediatrics, MaineHealth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MMP PEDIATRIC NEURO [11000028]
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Neonatal Encephalopathy
Keywords: Hypothermia, Induced; Telemedicine; Hospitals, Community
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telemedicine (Experimental): Babies that received telemedicine consult intervention.
  Interventions: Diagnostic Test: Telemedicine consult

INTERVENTIONS:
Diagnostic Test: Telemedicine consult — Utilizing telemedicine in community hospital for earlier identification of symptoms of neonatal encephalopathy.

SUMMARY:
This pilot intervention trial will assess the feasibility of a live consultation between community hospital providers and tertiary care providers employing a novel teleconsult platform, Maine Neonatal Encephalopathy Teleconsult (Maine NET), on the time to initiation of therapeutic hypothermia (TH) for 35 infants born in community hospitals in Maine compared with matched historical controls. Community hospital providers and tertiary care center provider satisfaction with the Maine NET platform will also be assessed. The hypothesis is that immediately available expert assessment via a teleconsult platform will promote earlier implementation of TH and be associated with high levels of provider satisfaction.

DETAILED DESCRIPTION:
The study will recruit a total of 125 infants from the participating centers and anticipate that 35 of these subjects will be treated with therapeutic hypothermia and be utilized for the comparative analysis to historical controls. Not all infants recruited and provided a Maine NET consultation will be treated with TH and to have an adequate sample size to make statistical comparisons with historical controls we need to enroll more than 35 participants to ensure 35 have been treated with TH for the comparative analysis.

In a secondary qualitative study, clinicians who completed Maine NET consults through the above clinical trial were interviewed about their experience with the consult. This secondary study will recruit up to 20 clinicians who completed a consult in this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

Infants included in this study will be born at a community hospital, will be in either high or moderate risk, will be younger than 6 hours of age at the time of the consultation and the decision will have been made to treat with TH. High risk infants will be defined as an umbilical cord pH of less than or equal to 7.0 or 5 minute APGAR score of less than or equal to 5 or a need for resuscitation (including respiratory support or chest compressions) or an abnormal exam (which may include flaccid tone, poor suck reflex or poor response to stimulation) or seizures at less than 6 hours of life. Moderate risk infants will be defined as an umbilical cord pH of less than or equal to 7.2 but greater than 7.0 or 5 minute APGAR score of less than 7 but greater than 5 or a perinatal event (such as placental abruption, uterine rupture, cord prolapse, or fetal-maternal hemorrhage) or an abnormal exam (which may include a hyper-alert state).

Exclusion Criteria:

Infants older than 6 hours at the time Maine NET is requested and infants for whom TH is not an appropriate therapy (e.g. due to premature birth or moribund status) will be excluded.

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 115 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexa Craig, MD, Principal Investigator — MaineHealth
Locations (1):
- Maine Medical Center, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Telemedicine
Started | 115
Completed | 115
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Telemedicine
Number analyzed (Participants) | 115
Age, Customized [Count of Participants; unit: Participants]
  0-6 hours | 115
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 101
  Unknown or Not Reported | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 97
  More than one race | 2
  Unknown or Not Reported | 11
Region of Enrollment [Number; unit: participants]
  United States | 115

OUTCOME MEASURES:

1. Primary Outcome: Time to Initiation of Therapeutic Hypothermia
Description: Time to initiation of therapeutic hypothermia
Time Frame: First 6 hours of life
Measure: Mean (Inter-Quartile Range); unit: hours
Arm/Group | Telemedicine
Number analyzed (Participants) | 113
hours | 4.5 [3.5 to 5.0]

ADVERSE EVENTS:
Time Frame: Duration of the telemedicine consultation (10-30 minutes)
Description: Adverse events were collected on patients during the duration of telemedicine consultation (time on consultation varied due to length of consent discussion if parent/guardian(s) had questions, patient acuity, and time for exam). This time period lasted for 10-30 minutes in duration and occurred within the first 6 hours of the child's life.
Arm/Group | Telemedicine
All-Cause Mortality (participants affected / at risk) | 0/113
Serious Adverse Events (participants affected / at risk) | 0/113
Other Adverse Events (participants affected / at risk) | 0/113

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT03706417/Prot_SAP_000.pdf